CLINICAL TRIAL: NCT07377695
Title: Comparison of Remimazolam Consumption According to Administration Method in Patients Undergoing Cerebrovascular Bypass Surgery: A Prospective Randomized Trial
Brief Title: Remimazolam Consumption: TCI vs. Manual Infusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Bypass-TCI
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Transcobalamins; remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCI (Experimental): Remimazolam administered via TCI (target Ce 0.7 μg/mL)
  Interventions: Other: Target-Controlled Infusion (TCI) of Remimazolam
- Manual Infusion (Active Comparator): Remimazolam administered via manual infusion (6 mg/kg/hr for induction, 1-2 mg/kg/hr for maintenance)
  Interventions: Other: Manual Infusion of Remimazolam

INTERVENTIONS:
Other: Target-Controlled Infusion (TCI) of Remimazolam — Remimazolam is administered using a target-controlled infusion (TCI) pump based on the Schuttler pharmacokinetic model. The initial target effect-site concentration (Ce) is set at 0.7 μg/mL and adjusted in 0.1 μg/mL increments to maintain a depth of anesthesia between Patient State Index (PSi) 25 and 50.
  Arms: TCI
Other: Manual Infusion of Remimazolam — Remimazolam is administered via traditional manual weight-based infusion. For anesthesia induction, a rate of 6 mg/kg/hr is used. For maintenance, the infusion rate starts at 1 mg/kg/hr and is adjusted in 0.2 mg/kg/hr increments to maintain a PSi between 25 and 50.
  Arms: Manual Infusion

SUMMARY:
The purpose of this prospective randomized controlled trial is to compare the total consumption of remimazolam between two different administration methods-Target-Controlled Infusion (TCI) and manual infusion-in patients undergoing cerebrovascular bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo cerebrovascular bypass surgery under general anesthesia.
* American Society of Anesthesiologists (ASA) Physical Status 1, 2, or 3
* Adults aged 19 years or older
* Patients who have provided prior written informed consent to participate in the study

Exclusion Criteria:

* Patients who do not consent to participate in the research
* Patients classified as ASA Physical Status 4
* Patients with a BMI ≤18.5 kg/m2 or 35.0 ≥ kg/m2
* History of allergy to benzodiazepine-class medications
* Patients with acute narrow-angle glaucoma
* Patients in a state of shock or coma
* Acute alcohol intoxication with suppressed vital signs , or patients with alcohol or drug dependency
* Presence of Sleep Apnea Syndrome or severe/acute respiratory failure
* Patients with lactose intolerance or hypersensitivity to Dextran 40

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Consumption of Remimazolam | From the start of anesthesia induction to the end of surgery (intraoperative period).
  The total cumulative dose of remimazolam ($mg$) administered from the initiation of anesthesia induction until the completion of the surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No